CLINICAL TRIAL: NCT02762240
Title: The Effectiveness of a Nationwide Mandatory Accreditation in General Practice in Denmark: A Randomized Controlled Trial
Brief Title: The Effectiveness of a Nationwide Mandatory Accreditation in General Practice in Denmark
Acronym: ACIAP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Southern Denmark (Other)
Collaborators: University of Copenhagen (Other); University of Aarhus (Other); The Danish Institute for Quality and Accreditation in Healthcare (Unknown)
Responsible Party: Principal Investigator, Frans Boch Waldorff, Professor, University of Southern Denmark
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: NAGEP_RCT01
Record Dates: First submitted 2016-03-29; First posted 2016-05-04 (Estimated); Last update posted 2016-05-26 (Estimated); Status verified 2016-05

CONDITIONS: Quality Control
Keywords: Accreditation; Certification; General Practice; Family Medicine; Randomized Controlled Trial
MeSH Terms: interventions — Early Intervention, Educational

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- DHQP 2016 (Active Comparator): This group consists of general practices allocated to undergo accreditation scheme in 2016.
  Interventions: Other: DHQP 2016
- DHQP 2018 (Placebo Comparator): This group consists of general practices allocated to undergo accreditation scheme in 2018.
  Interventions: Other: DHQP 2018

INTERVENTIONS:
Other: DHQP 2016 — DHQP for general practice consists of 16 standards with associated indicators within the following areas: 1. Quality and patient safety, 2. Patient safety critical standards, 3. Good patient continuity of care, 4. Management and organisation.
  Other Names: Early Intervention
  Arms: DHQP 2016
Other: DHQP 2018 — DHQP for general practice consists of 16 standards with associated indicators within the following areas: 1. Quality and patient safety, 2. Patient safety critical standards, 3. Good patient continuity of care, 4. Management and organisation.
  Other Names: Late Intervention
  Arms: DHQP 2018

SUMMARY:
Accreditation is used increasingly in health systems worldwide. However, there is a lack of evidence of the effectiveness of accreditation. The overall aim of this study is to evaluate the effectiveness of a mandatory accreditation in general practice.

DETAILED DESCRIPTION:
Accreditation has become a widespread tool for quality control and development, and large resources are spent upon development and implementation of accreditation systems in health care systems all over the world. Accreditation of healthcare systems has met some critique. Evidence for positive effects of accreditation has been called for, and health care professionals have expressed concerns about extra hours imposed by accreditation. However, only few studies have evaluated the effects of accreditation on central items, such as clinical outcomes and patient satisfaction. In general, the results from the different types of studies are ambiguous and there are only few well-accomplished effect studies. Hence, only two effect studies met the methodological inclusion criteria of a recent Cochrane review. None of these studies treated general practice. A review regarding status of accreditation in primary care concluded that there is a dearth of research on the nature and uptake of accreditation in this sector along with how accreditation affects outcomes of care, and whether it is an effective method to improve quality, perceptions of care, healthcare utilisation and costs. Two studies provided evidence to suggest that accreditation status was associated with infection control procedures, risk management programmes and quality improvement activities and after-treatment plans. However, in the latter case, post hoc analysis revealed that accreditation was associated with units' organizational contexts and referral sources as well as the nature of the competitive environment. The authors concluded that accreditation and licensing might reveal as much about a care units' institutional environments as about the quality of treatment provided. Accreditation is a relatively new instrument in general practice and its effects on clinical outcomes, patient satisfaction, general practitioners' (GPs') job satisfaction and organisational aspects must be evaluated in order to assess the overall utility for patients and society. Although accreditation has been implemented in general practice in nine European countries, and in Australia and New Zealand, research elucidating the effects of accreditation in general practice system, is strongly needed. In spite of this lack of evidence for effect of accreditation on clinical and patient related objectives, it has been decided to implement accreditation as a mandatory instrument in Danish general practice.

The Danish Healthcare Quality Programme (DHQP) is based on general principles for accreditation. The model contains a set of accreditation standards as well as an accreditation process. Accreditation has for a longer time period been mandatory in the secondary healthcare system in Denmark, and it has now been decided to include general practice as well. Hence, the DHQP has been adjusted to general practice. DHQP for general practice consists of 16 standards with associated indicators within the following areas: 1. Quality and patient safety, 2. Patient safety critical standards, 3. Good patient continuity of care, 4. Management and organisation. The first practices are accredited in January 2016, and at the end of 2018 all Danish practices should be accredited. An exception is practices with expected termination within 5 years.

Since accreditation is a complex intervention, containing several dimensions and active components, it is of great importance to elucidate these processes and mechanisms that become evident with the roll-out and implementation of accreditation and to examine the possible impact, accreditation may have on health care within primary care.

ELIGIBILITY:
Inclusion Criteria:

* General practices working under the Danish Health Insurance at June 2014

Exclusion Criteria:

* None

Max Age: 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1900 (Estimated)
Dates: Start 2014-06; Primary Completion 2017-07 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Changes in number of prescribed drugs in patients above 65 years in the observation periods. | 6 months periods
  Data regarding Prescription medication is retrieved from Nationwide Medication Database (MD)

SECONDARY OUTCOMES:
• Changes in the proportion of polypharmacy patients above 65 years (>5 prescribed drugs) between periods. | 6 months periods
  More than 5 prescribed drugs based on nationwide Medication Database (MD)
• Changes in Daily Drug Dose of NSAID without Proton-pump inhibitor in period between periods. | 6 months periods
  Based on nationwide Medication Database (MD)
• Changes in Daily Drug Dose of sleeping medicine between periods. | 6 month periods
  Based on nationwide Medication Database (MD)
Changes in the proportion of elderly above 75 receiving a preventive home visit between periods. | 6 month periods
  The regional practice remuneration system (RPRS)
Changes in the number of annual controls for chronic diseases between periods. | 6 month periods
  The regional practice remuneration system (RPRS)
Changes in the number of spirometry between periods | 6 month periods
  The regional practice remuneration system (RPRS)
Changes in proportion of practices with a reported adverse event between periods. | 6 month periods
  Danish Patient Security Database (DPSD)
Changes in the proportion of practices with a patient satisfaction survey between periods. | 6 month period
  Danish Patients Evaluation Practice database
Changes in mortality rates between periods. | 2 month periods from index date
  Statistics Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kirstine Andersen M, Pedersen LB, Waldorff FB. Retirement, job satisfaction and attitudes towards mandatory accreditation: a Danish survey study in general practice. BMJ Open. 2018 Aug 13;8(8):e020419. doi: 10.1136/bmjopen-2017-020419. PMID 30104311
- [Derived] Andersen MK, Pedersen LB, Siersma V, Bro F, Reventlow S, Sondergaard J, Kousgaard MB, Waldorff FB. Accreditation in general practice in Denmark: study protocol for a cluster-randomized controlled trial. Trials. 2017 Feb 13;18(1):69. doi: 10.1186/s13063-017-1818-6. PMID 28193288
- See also: Webpage of the Research group — http://www.akiap.dk